CLINICAL TRIAL: NCT04039022
Title: An Open-Label Study to Assess the Long-term Safety and Efficacy of AXS-05 in Subjects With Major Depressive Disorder
Brief Title: Open-Label Safety Study of AXS-05 in Subjects With Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXS-05-303
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression; Depression
Keywords: Depression; AXS-05; Dextromethorphan; Bupropion; Dopamine Reuptake Inhibitor; NMDA Receptor Antagonist; Nicotinic Acetylcholine Receptor Antagonist; Serotonin Reuptake Inhibitor; Axsome Therapeutics; Norepinephrine Reuptake Inhibitor; Sigma-1 Receptor Agonist; Glutamate Modulator; Antidepressant
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression | interventions — Dextromethorphan; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AXS-05 (Experimental)
  Interventions: Drug: AXS-05 (dextromethorphan and bupropion) oral tablets

INTERVENTIONS:
Drug: AXS-05 (dextromethorphan and bupropion) oral tablets — Oral tablets, taken twice daily for up to 12 months.

SUMMARY:
An open-label, long-term, safety study of AXS-05 in patients with major depressive disorder (MDD), including treatment resistant depression.

DETAILED DESCRIPTION:
A multi-center, open-label, long-term study to evaluate the safety and efficacy of AXS-05 in patients with major depressive disorder, including treatment resistant depression, treated for up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder, including treatment resistant depression
* Body mass index (BMI) between 18 and 40 kg/m^2, inclusive
* Agree to use adequate method of contraception for the duration of the study
* Additional criteria may apply

Exclusion Criteria:

* Suicide risk
* Pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study
* Additional criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (49):
  - Clinical Research Site, Phoenix, Arizona
  - Clinical Research Site, Little Rock, Arkansas
  - Clinical Research Site, Bellflower, California
  - Clinical Research Site, Beverly Hills, California
  - Clinical Research Site, Culver City, California
  - Clinical Research Site, Garden Grove, California
  - Clinical Research Site, Oakland, California
  - Clinical Research Site, Oceanside, California
  - Clinical Research Site, Panorama City, California
  - Clinical Research Site, Redlands, California
  - Clinical Research Site, San Diego, California
  - Clinical Research Site, Sherman Oaks, California
  - Clinical Research Site, Upland, California
  - Clinical Research Site, Cromwell, Connecticut
  - Clinical Research Site, Coral Springs, Florida
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site, Hollywood, Florida
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Lauderhill, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, North Miami, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Atlanta, Georgia
  - Clinical Research Site, Boise, Idaho
  - Clinical Research Site, Chicago, Illinois
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Las Vegas, Nevada
  - Clinical Research Site, Berlin, New Jersey
  - Clinical Research Site, Cherry Hill, New Jersey
  - Clinical Research Site, Toms River, New Jersey
  - Clinical Research Site, Jamaica, New York
  - Clinical Research Site, Rochester, New York
  - Clinical Research Site, Staten Island, New York
  - Clinical Research Site, Hickory, North Carolina
  - Clinical Research Site, Raleigh, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Middleburg Heights, Ohio
  - Clinical Research Site, Oklahoma City, Oklahoma
  - Clinical Research Site, Media, Pennsylvania
  - Clinical Research Site, Philadelphia, Pennsylvania
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, Dallas, Texas
  - Clinical Research Site, Fort Worth, Texas
  - Clinical Research Site, Houston, Texas
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, Wichita Falls, Texas
  - Clinical Research Site, Bellevue, Washington
  - Clinical Research Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AXS-05: AXS-05: Oral tablets, taken twice daily for up to 12 months.
Period: Overall Study
Arm/Group | AXS-05
Started | 876
Completed | 53
Not Completed | 823

BASELINE CHARACTERISTICS:
Population: Overall Safety Population (all subjects who received at least 1 dose of AXS-05)
Arm/Group | AXS-05
Number analyzed (Participants) | 876
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 560
  Male | 316
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 301
  White | 509
  More than one race | 10
  Unknown or Not Reported | 20

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent AEs (TEAEs) Following Dosing With AXS-05
Description: Types and rates of adverse events
Time Frame: Up to 12 months
Population: Primary Safety Population (subjects who continued beyond Week 6 of the trial)
Measure: Count of Participants; unit: Participants
Arm/Group | AXS-05
Number analyzed (Participants) | 707
Participants | 505

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were AEs with an onset date on or after the date of first dose. TEAEs were collected through 30 days after the last study visit.
Description: Overall Safety Population (all subjects who received at least 1 dose of AXS-05)
Arm/Group | AXS-05
All-Cause Mortality (participants affected / at risk) | 2/876
Serious Adverse Events (participants affected / at risk) | 21/876
Other Adverse Events (participants affected / at risk) | 609/876
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-05 (N=876)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-05 (N=876)
Dizziness (Nervous system disorders) | 111 (117)
Nausea (Gastrointestinal disorders) | 104 (110)
Headache (Nervous system disorders) | 77 (84)
Dry mouth (Gastrointestinal disorders) | 62 (64)
Decreased appetite (Metabolism and nutrition disorders) | 53 (53)
Constipation (Gastrointestinal disorders) | 29 (29)
Diarrhea (Gastrointestinal disorders) | 33 (37)
Nasopharyngitis (Infections and infestations) | 39 (41)
Upper respiratory tract infection (Infections and infestations) | 35 (42)
Somnolence (Nervous system disorders) | 30 (33)
Anxiety (Psychiatric disorders) | 34 (36)
Insomnia (Psychiatric disorders) | 31 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT04039022/Prot_SAP_000.pdf